CLINICAL TRIAL: NCT07025616
Title: Effectiveness of Buteyko Breathing Exercise in Children With Uncontrolled Asthma: A Single Blind, Randomized Controlled Trial
Brief Title: Effects of Buteyko Breathing Exercise in Children With Uncontrolled Asthma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ivan Sofian Wibowo (Other)
Collaborators: Fakultas Kedokteran Universitas Indonesia (Other); Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Sponsor-Investigator, Ivan Sofian Wibowo, dr., Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-07-1177
Record Dates: First submitted 2025-06-08; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Breathing Techniques; Asthma Control Level; Asthma in Children; Asthma Patients; Breathing Exercise
Keywords: Asthma; Buteyko; breathing retraining; pediatrics
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buteyko (Experimental): Buteyko breathing exercise plus pharmacological treatment
  Interventions: Behavioral: Buteyko; Drug: Asthma reliever and controller
- Control (Active Comparator): Pharmacological treatment
  Interventions: Drug: Asthma reliever and controller

INTERVENTIONS:
Behavioral: Buteyko — The Buteyko breathing exercise is a method that encourages nasal breathing, reducing breathing volume, and using breath-holding exercises to normalize breathing pattern
  Arms: Buteyko
Drug: Asthma reliever and controller — Asthma reliever and controller according to GINA (Global Initiative for Asthma) guideline

SUMMARY:
This randomized controlled trial study aimed to measure the effectiveness of the combination of 4-weeks Buteyko breathing exercises and pharmacological therapy compared with pharmacological therapy alone in children with uncontrolled asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 7-17 years
2. Uncontrolled or partially controlled asthma (GINA Symptom Control Tool score > 1)
3. Receive bronchodilator therapy, either oral or inhaler from a pediatrician.
4. Children and parents/care givers agree to participate in the study until the end, and parents/care givers sign the informed consent form.
5. Can understand instructions.

Exclusion Criteria:

1. Inpatients
2. Have received Buteyko breathing exercises or other breathing exercises.
3. Have congenital heart disease, pneumonia, or other significant and uncontrolled health disorders.
4. Have severe physical disabilities or mental retardation that could potentially prevent the implementation of Buteyko breathing exercises.
5. Have contraindications for spirometry examination

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Asthma control | At enrollment and end of fourth-week
  Level of asthma control measured by Asthma Control Questionnaire (ACQ) - Indonesian version.
  Minimum value 0, maximum value 6. Higher score means worse outcome.

SECONDARY OUTCOMES:
Asthma Quality of Life | At enrollment and end of fourth-week
  Measured by Pediatric Asthma Quality of Life Questionnaire standardized version (PAQLQ(S)) - Indonesian version.
  Minimum value 1, maximum value 7. Higher scores means better outcome.
Bronchodilator use | At end of fourth-week
  Bronchodilator use measured by logbook, recorded by caregiver of patients
FEV1 | At enrollment and end of fourth-week
  Forced Expiratory Volume in one second reflects degree of airway obstruction. Measured by spirometry.
FVC | At enrollment and end of fourth-week
  Forced Vital Capacity is total volume of air that can forcefully exhale after taking the deepest possible breath. Measured by spirometry.
FEV1/FVC | At enrollment and end of fourth-week
  Ratio of Forced Expiratory Volume in 1 second (FEV₁) to the Forced Vital Capacity (FVC). Measured by spirometry.
PEFR | At enrollment and end of fourth-week
  Peak Expiratory Flow Rate is maximum speed (flow rate) of air that can be blowed out in a single forced breath. Measured by spirometry.
Control Pause | At enrollment and end of fourth-week
  Duration of control pause

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Indonesia, Faculty of Medicine, Jakarta Pusat, Dki Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided